CLINICAL TRIAL: NCT05870917
Title: A Prospective, Single-center, Phase II Study of VRD-based Regimen Combined With CART-ASCT-CART2 Treatment in Patients With Newly Diagosed Primary Plasma Cell Leukemia
Brief Title: A Study of VRD-based Regimen Combined With CART-ASCT-CART2 Treatment in Patients With Primary Plasma Cell Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Gang An, Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Science & Peking Union Medical College, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAC-PPCL-001
Record Dates: First submitted 2023-04-29; First posted 2023-05-23 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Plasma Cell Leukemia
MeSH Terms: conditions — Leukemia, Plasma Cell | interventions — Bortezomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- VRD-based regimen Combined CART-ASCT-CART2 (Experimental): VRD：Bortezomib, Lenalidomide and Dexamethasone Bortezomib SC 1.3mg/sqm on day 1,8,15,22, Lenalidomide oral 25 mg on day 1-21, and Dexamethasone 40mg on day 1,8,15,22 in a 28-day cycle. Autologous BCMA-directed CAR-T cells, Double infusion intravenously at a target dose of (2-4)±20％ x 10^6 anti-BCMA CAR+T cells/kg respectively.
  Participants will receive VRD-based induction, first CAR-T infusion, VR consolidation, ASCT followed by the second CAR-T infusion, and R maintenance.
  Interventions: Biological: anti-BCMA CAR-T

INTERVENTIONS:
Biological: anti-BCMA CAR-T — Autologous BCMA-directed CAR-T cells, the double infusion intravenously at a target dose of (2-4)±20％ x 10^6 anti-BCMA CAR+T cells/kg respectively
  Other Names: Bortezomib, Lenalidomide and Dexamethasone

SUMMARY:
This is a single-arm, open-label study to evaluate the efficacy and safety of VRD-based Regimen (Bortezomib, Lenalidomide and Dexamethasone) combined with CART-ASCT-CART2 in Chinese patients with newly diagnosed primary plasma cell leukemia.

DETAILED DESCRIPTION:
The study is a prospective, single-arm, single-centre, phase II study designed to evaluate the efficacy and safety of treatment with VRD-based Regimen (Bortezomib, Lenalidomide and Dexamethasone) in combination with CART-ASCT-CART2 in Chinese patients with newly diagnosed primary plasma cell leukemia. Patients receive 3 cycles of induction therapy with VRD-based regimen followed by the first infusion of CAR-T cells. Patients then received 3 cycles of VR-based consolidation therapy, followed by ASCT and the second infusion of CAR-T cells. And R or R maintenance starts on day 100 after ASCT.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
2. Age ≥ 18 years and ≤ 65 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
4. Life expectancy at least 3 months
5. Definitive diagnosis of pPCL: meet the diagnosis criteria of multiple myeloma (refer to the Chinese guidelines for the diagnosis and management of multiple myeloma (revised 2022) criteria) and meeting any of the following:

   1. the proportion of tumor plasma cells in peripheral blood leukocytes ≥ 5%;
   2. absolute value of peripheral blood tumorigenic plasma cells exceeds 2×10^9/L.
6. Patients have not received previous anti-myeloma related therapy.
7. Measurable disease, as defined by at lease one of the following:

   1. Serum monoclonal paraprotein (M-protein) level ≥5g/L.
   2. urine M-protein level ≥200 mg/24 hours.
   3. If the serum and urine M-protein are unmeasurable, abnormal serum free light chain (FLC) ratio and affected FLC ≥10 mg/dL.
8. Bone marrow sample is confirmed as BCMA-positive by flow cytometry or pathological examination.
9. Routine blood tests (performed within 7 days, no RBC transfusion, no G-CSF/GM-CSF/platelet agonists, no drug correction within 14 days before screening, no PLT transfusion within 7 days) : ANC ≥ 1.0 x 10^9/L, PLT ≥ 50 x 10^9/L.
10. All screening blood biochemistry: tests should be performed according to the protocol and within 14 days before enrollment. Screening laboratory values must meet the following criteria:

    1. Total bilirubin<1.5 x upper limit of normal (ULN);
    2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST);
    3. Creatinine clearance ≥ 50mL/min (calculated using Cockroft-Gault formula).
11. Patients must be able to take prophylactic anticoagulant therapy as recommended by the study.
12. The woman is not breastfeeding, is not pregnant and agrees not to be pregnant during the study period and for the following 12 months. Male patients agreed that their spouse would not become pregnant during the study period and for 12 months thereafter.
13. Willing and able to complete the study procedures and follow-up examinations.

Exclusion Criteria:

1. Secondary plasma cell leukemia.
2. With central nervous system (CNS) involvement.
3. Ineligible for autologous stem cell transplantation, such as severe cardiopulmonary disorders.
4. Known intolerant, allergic, or resistant to glucocorticoids, bortezomib, lenalidomide, Venetoclax, Selinexor and BCMA-CART cellular products.
5. Patients had major surgery within 2 weeks before randomization (for example, general anesthesia), or is not fully recovered from the surgery, or surgery is arranged during study period.
6. Patients with unstable or active cardiovascular system disease, meeting any of the following:

   1. Unstable angina pectoris, symptomatic myocardial ischaemia, myocardial infarction or coronary artery reconstruction within 180 days prior to the first dose.
   2. Uncontrolled hypertension (>140/90 mmHg with blood pressure fluctuations of more than 180/100 mmHg over a 6-month period).
   3. Uncontrolled and clinically significant conduction abnormalities (e.g. patients with ventricular arrhythmias controlled by antiarrhythmic medication), not excluding patients with 1st degree atrioventricular (AV) block or asymptomatic left anterior bundle branch block/right bundle branch block (LAFB/RBBB)).
   4. Congestive heart failure (CHF) classification ≥ grade 3 as defined by the New York Heart Association (NYHA).
   5. Left ventricular ejection fraction (LVEF) <50% on echocardiography.
   6. History of stroke or intracranial haemorrhage within 12 months prior to screening.
   7. Presence of a serious thrombotic event prior to treatment.
7. Known positive serology for HIV or HIV seropositivity.
8. Active hepatitis B or C infection. Screening requires serologic testing for hepatitis. If hepatitis B surface antigen and hepatitis B core antibody were positive, a negative DNA polymerase chain reaction (PCR) result was needed before enrollment (after anti-hepatitis B therapy, a negative DNA polymerase PCR result was confirmed before enrollment). If the hepatitis C antibody was positive, the RNA PCR test should be negative prior to enrollment.
9. Ongoing active infection.
10. Prior history of malignancies, unless free of the disease for ≥ 5 years.
11. Pregnant or breast feeding females.
12. Any active gastrointestinal dysfunction that affects the patient's ability to swallow tablets, or any active gastrointestinal dysfunction that may affect the absorption of the studied treatment medication.
13. According to the researcher's judgment, any condition including but not limited to serious mental illness, medical illness, or other symptoms/conditions that may affect study treatment, compliance, or the capability of providing informed consent.
14. Necessary medication or supportive therapy is contraindicated with study treatment.
15. Any other medical condition or comorbidity that might interfere with subject's participation.
16. Patients undergoing other experimental therapies.
17. Patients are not willing to or cannot comply with study scheme.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 2 year
  The incidence of treatment-emergent adverse events (TEAEs)
Overall response rate (ORR) | after induction therapy, 1 month after the first CAR-T cell transfusion, the consolidation therapy ends, 6 months after the second CAR-T cell transfusion
  ORR(including sCR / CR / VGPR / PR, based on IMWG criteria)
Progression free survival (PFS) | 1 year
  Is defined as time from first induction date to first documentation of PD, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Complete response rate (CRR) | after induction therapy, 1 month after the first CAR-T cell transfusion, the consolidation therapy ends, 6 months after the second CAR-T cell transfusion
  CR or better is defined as percentage of participants who achieve a CR response or Stringent Complete Response (sCR) response according to IMWG criteria
Overall survival (OS) | 1 year
  Is defined as time from first induction date to time of death due to any cause
MRD-negative Rate | after induction therapy, 1 month after the first CAR-T cell transfusion, the consolidation therapy ends, 6 months after the second CAR-T cell transfusion
  MRD negative by flow cytometry
Duration of Remission (DOR) | 2 year
  Duration from the first evaluation of at least partial remission (PR) to the onset of disease progression or death due to disease progression (whichever occurs first)

OTHER OUTCOMES:
The CART cell duration in vivo | 1 year
  The copies of BCMA-CART DNA in peripheral blood with qPCR method

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, China